CLINICAL TRIAL: NCT00268632
Title: A Multicenter Prospective Study to Assess the Impact of Physician's Reinforcement on the Subject's Compliance and Persistence on Treatment Using Feedback on Bone Markers in Previously Undiagnosed Postmenopausal Osteoporotic Women Treated With Risedronate.
Brief Title: IMPACT Study (Improving Measurements of Persistence on "ACtonel" Treatment)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4001
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

INTERVENTIONS:
Drug: risedronate

SUMMARY:
The primary objective of this study is to assess the impact of physician's reinforcement using bone marker data on the subject's compliance (at least 50% drug taken) and persistence on treatment after one year in postmenopausal osteoporotic women.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women,
* Caucasian, Oriental or Multiracial
* not previously diagnosed for osteoporosis.

Exclusion Criteria:

* Females of black descent and for the US african american are excluded because of the very low incidence of postmenopausal osteoporosis
* and having used oral or parenteral glucocorticoids (>= 5 mg prednisone or equivalent per day) within 3 months of starting study drug or for more than one month within six months prior to study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1999-08; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
To assess the impact of physician's reinforcement using bone marker data on the treatment adherence of women with PMO. | collected at week 10 and 22

SECONDARY OUTCOMES:
to establish the profile of the unrecognized osteoporotic woman (PVD-, RF-) using a risk factor questionnaire for osteoporosis | During the study conduct
to assess the decrease of type I collagen breakdown products(urinary NTX and serum CTX) | after 10 and 22 weeks of treatment
To assess the change in BMD of both total hip and lumbar spine; | at week 52 compared to baseline
osteoporosis-related genotyping. | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Lex van de Langerijt, Study Director — Sanofi

REFERENCES:
- [Result] Delmas PD, Vrijens B, Eastell R, Roux C, Pols HA, Ringe JD, Grauer A, Cahall D, Watts NB; Improving Measurements of Persistence on Actonel Treatment (IMPACT) Investigators. Effect of monitoring bone turnover markers on persistence with risedronate treatment of postmenopausal osteoporosis. J Clin Endocrinol Metab. 2007 Apr;92(4):1296-304. doi: 10.1210/jc.2006-1526. Epub 2007 Jan 23. PMID 17244788
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?db=pubmed&cmd=Retrieve&dopt=AbstractPlus&list_uids=17244788&query_hl=2&itool=pubmed_docsum